CLINICAL TRIAL: NCT05586022
Title: Risk Factors for Adverse Outcomes of Endovascular Revascularization in Lower Extremity Arteriosclerosis Occlusion: a Prospective Observational Study
Brief Title: Risk Factors for Adverse Outcomes of Endovascular Revascularization in Lower Extremity Arteriosclerosis Occlusion
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-346
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting 10 mL blood samples from participants are collected for the detection of blood biochemical indicators, such as myocardial enzymes, troponin, liver function, kidney function, blood lipids, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lower extremity arterial occlusion undergoing endovascular revascularization: We will enroll the patients with lower extremity arterial occlusive disease admitted to the Department of Vascular Surgery of The First Affiliated Hospital of Xi 'an Jiaotong University. These patients undergo successful endovascular revascularization of the diseased vessel.
  Interventions: Procedure: endovascular revascularization

INTERVENTIONS:
Procedure: endovascular revascularization — percutaneous balloon dilatation, stent implantation, plaque resection, laser plasty, cutting balloon, drug balloon, cryoballoplasty, thrombolytic therapy with drugs or thrombectomy

SUMMARY:
Arteriosclerosis obliterans (ASO) is one of the most common peripheral artery diseases (PADs) which causes ischemic symptoms of the lower limbs. Endovascular treatment has emerged as the most commonly used and efficient treatment option for PAD. However, adverse cardiovascular and lower extremity outcomes are inevitable, which remains a challenge for the vascular surgeon. ASO can be characterized by intermittent claudication, ischemic resting pain, and severe lower extremity ischemia. Known risk factors for lower extremity ASO include smoking, diabetes, hypertension, hyperlipidemia, hyperhomocysteinemia, chronic renal insufficiency, inflammatory indicators, etc.

Endovascular revascularization is widely used at present. Many clinical centers choose endovascular therapy as the revascularization method of choice because of the lower incidence of complications and mortality compared with surgery, and the possibility of switching to open surgery if treatment fails. Luminal therapy is recommended when intermittent claudication affects quality of life, exercise or medical therapy is not effective, and clinical features suggest that endovascular therapy can improve the patient's symptoms and has a good risk benefit. At present, endovascular revascularization is widely used, but the incidence of adverse cardiovascular and lower extremity outcomes is still high, and the risk factors affecting the adverse outcomes after endovascular revascularization are still unclear.

The aim of this study is to explore the risk factors affecting the poor outcome of endovascular revascularization for lower extremity ASO, and to provide precise prevention strategies for improving the prognosis of the patients. This study was designed as a single-center, prospective observational study. A total of 500 adult patients with lower extremity ASO who underwent endovascular revascularization in the Departments of Vascular Surgery and Peripheral Vascular in the First Affiliated Hospital of Xi'an Jiaotong University were enrolled as the study cohort. The exclusion criteria includes patients with severe infections, tumors, liver and kidney failure, autoimmune diseases, and incomplete baseline data. Demographic characteristics, comorbidities, and serum biochemical parameters were collected at baseline. The patients were followed up 1-3 years after interventional therapy. Follow-up included adverse cardiovascular events (cardiovascular death, acute myocardial infarction, stroke), lower extremity adverse events (resting pain, gangrene, amputation), and all-cause death. Multivariate COX regression analysis is used to analyze the influencing factors of poor prognosis in patients with lower extremity ASO undergoing endovascular revascularization.

DETAILED DESCRIPTION:
Arteriosclerosis obliterans (ASO) is one of the most common peripheral artery diseases (PADs) which causes ischemic symptoms of the lower limbs. Endovascular treatment has emerged as the most commonly used and efficient treatment option for PAD. However, adverse cardiovascular and lower extremity outcomes are inevitable, which remains a challenge for the vascular surgeon. Pathologically, stenosis of the lower extremity arteries caused by arteriosclerosis has been regarded as the main cause of PAD. Lower extremity ASO is a chronic progressive disease caused by arteriosclerosis, which causes thickening of the intima of the feeding arteries of the lower extremity, lumen stenosis or occlusion, and insufficient blood supply to the diseased limb, resulting in intermittent claudication of the lower extremity, decreased skin temperature, pain, and even ulceration or necrosis. It is often the manifestation of systemic arteriosclerosis vasculopathy in the lower extremity arteries. ASO can be characterized by intermittent claudication, ischemic resting pain, and severe lower extremity ischemia. The main cause of lower limb ASO is atherosclerosis, and its incidence rises with age. The incidence of ASO in people over 70 years old is 15-20%, and the incidence of ASO in men is slightly higher than that in women. Known risk factors for lower extremity ASO include smoking, diabetes, hypertension, hyperlipidemia, hyperhomocysteinemia, chronic renal insufficiency, inflammatory indicators, etc.

In terms of treatment, in addition to the treatment of cardiovascular risk factors such as lipid-lowering drugs, antihypertensive drugs, diabetes treatment, smoking cessation, antiplatelet and anticoagulant therapy, endovascular revascularization is widely used at present. Many clinical centers choose endovascular therapy as the revascularization method of choice because of the lower incidence of complications and mortality compared with surgery, and the possibility of switching to open surgery if treatment fails. Luminal therapy is recommended when intermittent claudication affects quality of life, exercise or medical therapy is not effective, and clinical features suggest that endovascular therapy can improve the patient's symptoms and has a good risk benefit. There are many endovascular techniques for the treatment of lower extremity ASO, including percutaneous balloon dilatation, stent implantation, plaque resection, laser plasty, cutting balloon, drug balloon, cryoballoplasty, thrombolytic therapy with drugs or thrombectomy. At present, endovascular revascularization is widely used, but the incidence of adverse cardiovascular and lower extremity outcomes is still high, and the risk factors affecting the adverse outcomes after endovascular revascularization are still unclear.

Therefore, the purpose of this study is to explore the risk factors affecting the poor outcome of endovascular revascularization for lower extremity ASO, and to provide precise prevention strategies for improving the prognosis of the patients. This study was designed as a single-center, prospective observational study. A total of 500 adult patients with lower extremity ASO who underwent endovascular revascularization in the Departments of Vascular Surgery and Peripheral Vascular in the First Affiliated Hospital of Xi 'an Jiaotong University were enrolled as the study cohort. The exclusion criteria includes patients with severe infections, tumors, liver and kidney failure, autoimmune diseases, and incomplete baseline data. Demographic characteristics, comorbidities, and serum biochemical parameters were collected before operation. The patients were followed up 1 year after operation. Follow-up included adverse cardiovascular events (cardiovascular death, acute myocardial infarction, stroke), lower extremity adverse events (resting pain, gangrene, amputation), and all-cause death. According to the estimation principle of multivariate COX regression for sample size, the minimum sample size of each group should be multiplied by the observed variable by 10-15, and the observed variable is estimated to be 10-15, so the minimum sample size of each group is estimated to be between 150-225, and the overall sample size is about 300. Multivariate COX regression analysis is used to analyze the influencing factors of poor prognosis in patients with lower extremity ASO undergoing endovascular revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with lower extremity arterial occlusive disease who underwent successful endovascular revascularization.
* Preoperative baseline clinical data were complete.
* Patients who completed the informed consent form.

Exclusion Criteria:

* Patients with severe infections, tumors, liver and kidney failure, and autoimmune diseases.
* Patients with incomplete baseline data.
* Patients lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included adult patients with lower extremity arterial occlusive disease who had successfully undergone endovascular revascularization in the First Affiliated Hospital of Xi 'an Jiaotong University. These patients had complete preoperative baseline data including demographic characteristics, comorbidities, and related blood biochemical indicators, and signed informed consent to accept follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
adverse cardiovascular events | Patients were followed up from the day of endovascular revascularization to 1 year after operation
  cardiovascular death, acute myocardial infarction, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Qingbin Zhao, Doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No